CLINICAL TRIAL: NCT01321684
Title: The Effect of Spinal Flexion in the Lateral Decubitus Position on the Unilaterality During Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1006-100-322
Record Dates: First submitted 2011-03-18; First posted 2011-03-23 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Spinal Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: lateral decubitus position with full spinal flexion — The patients maintained the lateral decubitus position with the hips and back fully flexed for 15 minutes.
Other: lateral decubitus position without spinal flexion — the patients are allowed to straighten their flexed hips and back to obtain the normal lordotic curvature of spinal column

SUMMARY:
For unilateral spinal block, spinal local anesthetics should take effect on the spinal nerves of one side. With full flexion of the spine, the cauda equina becomes tightened and hangs in the middle of the subarachnoid space. This study was performed to assess if flexion of the vertebral column facilitates unilateral spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status Ⅰ-Ⅱ, scheduled for elective knee arthroscopy under spinal anesthesia

Exclusion Criteria:

* Hemodynamically unstable patients
* Lumbar disease
* patients with back pain

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Time for the complete regression of pinprick spinal analgesia on the nondependent legs | Sensory and motor blockade were evaluated within 3 hour of intrathecal injection

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university hospital, Seoul, South Korea